CLINICAL TRIAL: NCT01252108
Title: Phase 2A Open-label Study to Evaluate Safety, Tolerability, and Antimicrobial Activity of Single, Daily Doses of SQ109 in Urea Breath Test Positive Volunteers
Brief Title: Evaluation of SQ109 Plus PPI in Urea Breath Test-Positive Volunteers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Sequella, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SQ109-H001
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; peptic ulcer disease; stomach ulcers; gastric cancer
MeSH Terms: conditions — Peptic Ulcer; Stomach Ulcer; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): All subjects receive SQ109
  Interventions: Drug: SQ109

INTERVENTIONS:
Drug: SQ109 — 300 mg SQ109 daily for 14 days

SUMMARY:
Helicobacter pylori infection of the gastric epithelium is the most common bacterial infection worldwide. Its global prevalence is estimated at 50%, though the burden falls disproportionately on the developing world, where the prevalence in some areas is 80%. H. pylori infection is generally acquired during childhood, and without specific antibiotic treatment can persist for life. The infection is generally clinically asymptomatic during childhood, and even in adulthood 80-90% of infected individuals will remain asymptomatic (although they may transmit the bacteria).

SQ109 is a new, small molecule antibiotic with characteristics that make it particularly attractive to evaluate against H. pylori. In brief, SQ109 is orally bioavailable, acid-stable, has in vitro activity against H. pylori and achieves high intracellular concentration (which may be important to effect bacterial eradication).

Based on the antimicrobial activity and clinical safety, SQ109 will be evaluated in this clinical trial to assess safety and antimicrobial activity in adults infected with H. pylori. Data from this study will help determine whether larger safety and efficacy studies in individuals with H. pylori-associated duodenal ulcer disease are warranted.

DETAILED DESCRIPTION:
A total of 30 Urea Breath Test (UBT)-Positive volunteers will be enrolled. Each subject will receive SQ109 150 mg bid with PPI or 300 mg qd by mouth daily for 14 consecutive days.

Major Inclusion/Exclusion Criteria:

1. Subject must be 18 to 45 years of age (inclusive).
2. Subject must have 2 positive Urea Breath Tests (UBT) obtaining during screening, and no other clinically significant disease (i.e., hematology, clinical chemistry and urinalysis tests must be within study-defined ranges. Clinical tests must be performed within 14 days of receiving first dose of study drug.
3. Body Mass Index (BMI) must be between 18 and 33 kg/m2 inclusive.
4. Subject must be able to give voluntary written informed consent before any study related procedure is performed.

Objectives:

1. To determine the safety and tolerability of SQ109 administered daily for 14 consecutive days in male and female Urea Breath Test (UBT)-positive subjects.
2. To assess antimicrobial activity against H. pylori of SQ109 administered daily for 14 days in UBT-positive subjects.

Design: Each subject will undergo screening evaluations within 14 days of study entry (Day 1) and baseline evaluations Day -14 and Day -2 to Day 1 (up to 14 days prior to the first dose). On Day 1 (first day of dosing), the subject will be administered study drug and undergo the Day 1 procedures. Throughout the 14 days of treatment phase of the study each subject will be assessed daily for adverse events (AEs). Laboratory safety evaluations will be performed on Day 7, 8, 9, or 10, and on Day 14, and Day 21. On Days 1, 4, 7, 10, 14, 21, and 28 each subject will have a UBT. On Follow-up Days 21 and 28 each subject will return to the study unit to have safety assessments.

Outcome Measures:

Safety and tolerability will be evaluated by a review of physical examinations, neurological examinations, vital signs assessments, 12-lead ECGs, routine clinical laboratory tests (including chemistry and hematology data), and AE assessments.

Efficacy Outcome Measures consist of serial UBT assessments for evidence of H. pylori in the gastrointestinal tract collected at baseline, during the 14 days of SQ109 administration, and during the 14 day follow-up period.

ELIGIBILITY:
Major Inclusion Criteria:

1. Subject must be 18 to 45 years of age (inclusive).
2. Subject must have 2 positive Urea Breath Tests (UBT) obtaining during screening, and no other clinically significant disease (i.e., hematology, clinical chemistries and urinalysis tests must be within study-defined ranges (See Appendix B). Clinical tests must be performed within 14 days of receiving first dose of study drug.
3. Body Mass Index (BMI) must be between 18 and 30 kg/m2 inclusive.
4. Subject must be able to give voluntary written informed consent before any study related procedure is performed.
5. If female, has no childbearing potential or agrees to avoid becoming pregnant from the day of screening through their entire participation in the trial (Day 42) by using one of the following acceptable methods of birth control plus recommended use of a barrier method (condom) by the male partner (even if vasectomized):

   1. intrauterine contraceptive device; or
   2. diaphragm in combination with contraceptive jelly, cream, or foam; or
   3. spermicide; or
   4. abstinence.

Major Exclusion Criteria:

1. A history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition which would jeopardize the safety of the subject or impact the validity of the study results.
2. Abnormal diet during the 4 weeks preceding the study.
3. Use of any OTC or prescription medication, including vitamins and herbal supplements, within 7 days prior to Day 1 of the study, unless the substance would not likely impact on the conduct of this study.
4. Current medical condition (other than H. pylori infection) requiring treatment with medication, either prescription or OTC.
5. Treatment with any known CYP450 enzyme altering drugs such as azoles, antifungals, barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to Day 1 of the study.
6. Positive blood screen for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibody and/or a positive urine screen for alcohol or drugs of abuse.
7. Baseline QTc interval >450 msec (males) or >470 msec (females)or a family history of prolonged QTc syndrome or premature cardiac death.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Activity of SQ109 against H. pylori measured by Urea Breath Test Results | During the 14 days of drug adminstration and 14 days of follow-up
  In addition to assessment of safety and tolerability of SQ109, Preliminary efficacy will be assessed by serial Urea Breath Tests during the 14 days of drug administration, and recurrence will be assessed during the 14 days following the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lanza, MD, Principal Investigator — Houston Institue for Clinical Research